CLINICAL TRIAL: NCT00338013
Title: Patient Sleep Position Questionnaire
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Karen Joos, Associate Professor of Ophthalmology, Vanderbilt University
Other Study IDs: Vanderbilt IRB # 000832
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Sleep
Keywords: sleep

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
You are being asked to participate in this study because we would like to know if sleeping may affect eye pressure.

DETAILED DESCRIPTION:
Completion of the questionnaire is done solely for research purposes and is not part of your routine care.

Approximate duration- Up to 10 minutes to complete the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma
* Age-matched controls
* Adults

Exclusion Criteria:

* Medical students
* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2001-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Joos, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States